CLINICAL TRIAL: NCT05322798
Title: High-frequency Spinal Cord Stimulation in Treatment of Chronic Limb-Threatening Ischemia (HEAL-SCS): a Randomized Clinical Trial
Brief Title: High-frequency SCS in Treatment of Chronic Limb-Threatening Ischemia
Acronym: HEAL-SCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEAL-SCS
Record Dates: First submitted 2022-03-30; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Chronic Limb-Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HF-SCS (Experimental): SCS system implantation with high-frequency stimulation availability
  Interventions: Procedure: High-frequency SCS
- LF-SCS (Active Comparator): Conventional SCS system implantation
  Interventions: Procedure: Low-frequency SCS

INTERVENTIONS:
Procedure: High-frequency SCS — Continous high-frequency stimulation (frequency - 1kHz, pulse width - 30 µs).
  Arms: HF-SCS
Procedure: Low-frequency SCS — Continuous conventional stimulation (frequency - 30-60 Hz, pulse width - 250-500 µs).
  Arms: LF-SCS

SUMMARY:
The study of high-frequency spinal cord stimulation (SCS) efficacy in the treatment of chronic limb-threatening ischemia (CLTI)

DETAILED DESCRIPTION:
Open-label, parallel-group, randomized study with a 1:1 allocation ratio to check the hypothesis of whether high-frequency-SCS (HF-SCS) is better than conventional low-frequency (LF-SCS) for pain relief in patients with chronic limb-threatening ischemia (CLTI).

ELIGIBILITY:
Inclusion Criteria:

* non-reconstructable critical limb-threatening ischemia (CLTI)
* Fontaine stage IIB-IV
* VAS score 5/10 or more
* succesful SCS trial

Exclusion Criteria:

* intractable acute infection
* allergy to SCS component
* ulcerations larger than 3 cm2
* inadequate patient compliance
* life expectancy less than 12 months
* patient refuse to participate in any stage of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-08-12 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) score | 12 months
  score by visual analog scale (0-10)

SECONDARY OUTCOMES:
Visual analog scale (VAS) score | 3 months
  score by visual analog scale (0-10)
Walking Impairment Questionnaire (WIQ) - calf pain severity | 3 months
  walking impairment questionnaire score for calf pain severity (0-100)
Walking Impairment Questionnaire (WIQ) - calf pain severity | 12 months
  walking impairment questionnaire score for calf pain severity (0-100)
Walking Impairment Questionnaire (WIQ) - walking distance | 3 months
  walking impairment questionnaire score for walking distance (0-100)
Walking Impairment Questionnaire (WIQ) - walking distance | 12 months
  walking impairment questionnaire score for walking distance (0-100)
Walking Impairment Questionnaire (WIQ) - walking speed | 3 months
  walking impairment questionnaire score for walking speed (0-100)
Walking Impairment Questionnaire (WIQ) - walking speed | 12 months
  walking impairment questionnaire score for walking speed (0-100)
Walking Impairment Questionnaire (WIQ) - stair climbing | 3 months
  walking impairment questionnaire score for stair climbing (0-100)
Walking Impairment Questionnaire (WIQ) - stair climbing | 12 months
  walking impairment questionnaire score for stair climbing (0-100)
Short form 36 health survey (SF-36) - physical component summary | 3 months
  quality of life by physical component summary of short form 36 health survey (0-100)
Short form 36 health survey (SF-36) - physical component summary | 12 months
  quality of life by physical component summary of short form 36 health survey (0-100)
SF-36 - mental component summary | 3 months
  quality of life by mental component summary of short form 36 health survey (0-100)
SF-36 - mental component summary | 12 months
  quality of life by mental component summary of short form 36 health survey (0-100)
TcPO2 (rest) | 12 months
  transcutaneous oxygen tension at rest
TcPO2 (orthostatic probe) | 12 months
  transcutaneous oxygen tension during active orthostatic probe

CONTACTS AND LOCATIONS:
Overall Officials: Kiril Orlov, MD, PhD, Principal Investigator — Meshalkin National Medical Research Centre
Locations (1):
- Meshalkin National Medical Research Center, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilchukov M, Kiselev R, Gorbatykh A, Klinkova A, Murtazin V, Kamenskaya O, Orlov K. High-Frequency versus Low-Frequency Spinal Cord Stimulation in Treatment of Chronic Limb-Threatening Ischemia: Short-Term Results of a Randomized Trial. Stereotact Funct Neurosurg. 2023;101(1):1-11. doi: 10.1159/000527309. Epub 2023 Jan 6. PMID 36617410